CLINICAL TRIAL: NCT07056179
Title: REST Trial: Effects of a Brief Behavioral Intervention to Maintain Sleep Regularity in Young Adults Over the Christmas Break
Brief Title: Brief Behavioral Intervention to Maintain Sleep Regularity in Young Adults Over the Christmas Break
Acronym: REST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: The University of Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, YU Jucheng, Research Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20250606_REST; REC/24-25/0554 (Other: Hong Kong Baptist University)
Record Dates: First submitted 2025-07-07; First posted 2025-07-09 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Sleep
Keywords: sleep regularity; brief behavioral intervention; young adults

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants cannot be blinded. However, they will be unaware of the true aim of the study and will be informed that the intervention is intended to enhance overall well-being. Outcome measures will be administered by research personnel who are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief behavioural intervention group (Experimental): Participants will receive a brief behavioral intervention comprising a regularity-focused sleep diary, 10 tips for maintaining sleep regularity, and a sleep education information sheet. The regularity-focused sleep diary is designed to emphasize in-bed and out-of-bed times, drawing participants' attention to their sleep regularity. Participants will be provided with a yellow marker to highlight their sleep periods. The 10 tips for maintaining sleep regularity include establishing a consistent out-of-bed time, using natural light to regulate the circadian clock, adjusting mealtimes, etc. The sleep education sheet contains information on reducing caffeine intake in the afternoon, limiting screen time before bed, etc.
  Interventions: Behavioral: Brief behavioural intervention
- Health education control group (Placebo Comparator): Participants will receive general health information without specific emphasis on sleep, such as weight control, smoking cessation, etc.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Brief behavioural intervention — Participants will receive a brief behavioural intervention comprising a regularity-focused sleep diary, 10 tips for maintaining sleep regularity, and a sleep education information sheet. The regularity-focused sleep diary is designed to emphasize in-bed and out-of-bed times, drawing participants' attention to their sleep regularity. Participants will be provided with a yellow marker to highlight their sleep periods. The 10 tips for maintaining sleep regularity include establishing a consistent out-of-bed time, using natural light to regulate the circadian clock, adjusting mealtimes, etc. The sleep education sheet contains information on reducing caffeine intake in the afternoon, limiting screen time before bed, etc.
  Arms: Brief behavioural intervention group
Behavioral: Health education — Participants will receive general health information without specific emphasis on sleep, such as weight control, smoking cessation, etc.
  Arms: Health education control group

SUMMARY:
This study will employ a randomized controlled trial design to investigate the effects of a brief behavioral intervention that includes (1) self-recording of a regularity-focused sleep diary, (2) 10 strategies for maintaining sleep regularity, and (3) a sleep education information sheet on the maintenance of sleep regularity in young adults during the Christmas break.

ELIGIBILITY:
Inclusion Criteria:

1. Young adults aged 18-24 years;
2. Will stay in Hong Kong during the study period;
3. Will not engage in any activities that require a fixed sleep or wake-up time (e.g., work or study during the holiday period) as these activities could regularize the sleep schedule and potentially contaminate the results.

Exclusion Criteria:

1. Have been in a different time zone within two weeks before the baseline assessment;
2. Diagnosed with circadian rhythm disorders such as delayed sleep-wake phase disorder (DSWD), advanced sleep-wake phase disorder (ASWD), irregular sleep-wake rhythm disorder (ISWRD), and non-24-hour sleep-wake rhythm disorder (N24WSD);
3. Diagnosed with sleep disorders that directly/indirectly interfere with sleep regularity (e.g., insomnia, sleep apnea);
4. Use of medications or treatment that may influence sleep regularity (e.g., hypnotics, antidepressants);
5. Diagnosed with serious physical or mental diseases such as cancer, end-stage liver or kidney diseases, schizophrenia, and psychosis.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Sleep regularity | From baseline assessment to the end of intervention at 3 weeks
  Sleep regularity will be measured by the validated Chinese version of sleep regularity questionnaire (SRQ), which shows excellent reliability and validity. SRQ consists of six items focusing on two dimensions, circadian regularity and sleep continuity regularity. Each item is rated on a scale ranging from 0 (not at all) to 4 (very much) in terms of the degree to which they agreed with each statement, with higher scores indicating higher sleep regularity.

SECONDARY OUTCOMES:
Severity of depression | From baseline assessment to the end of intervention at 3 weeks
  The severity of depression will be measured by the Patient Health Questionnaire - 9 item (PHQ-9). It asks participants how often they experienced depressive symptoms over the past 2 weeks. PHQ-9 comprises 5 categories: 0-4 indicates minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, and ≥20 severe depression.
Severity of anxiety | From baseline assessment to the end of intervention at 3 weeks
  The severity of anxiety will be measured by the Generalized Anxiety Disorder - 7 item (GAD-7). The cut-off scores of GAD-7 are: 0-4 indicates minimal anxiety, 5-9 mild anxiety, 10-14 moderate anxiety, and ≥15 severe anxiety.
Work and social functioning | From baseline assessment to the end of intervention at 3 weeks
  Work and social functioning will be assessed using the Work and Social Adjustment Scale (WSAS), a 5-item instrument in which each item is rated on a 9-point Likert scale (0 = not at all, 8 = very severely). The total WSAS score ranges from 0 to 40, with lower scores indicating better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Danny YU, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Hong Kong Baptist University, Kowloon City, Kowloon Tong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan, and analytic code will be deposited in an open registry when the study is published.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will be available after the publication of the main results for 3 years.
Access Criteria: Study protocol, statistical analysis plan, and analytic code will be deposited in an open registry when the study is published for academic use only.